CLINICAL TRIAL: NCT05444907
Title: Understanding Deep Brain Stimulation-induced Mania: Finding Potential Predictors to Optimize Treatment
Brief Title: Deep Brain Stimulation-Induced Mania in Parkinson's Disease
Acronym: BPD_DBS
Status: Recruiting | Type: Observational
Sponsor: Albino Maia (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental (Other Government); Centro Hospitalar De São João, E.P.E. (Other); Unidade Local de Saúde de Coimbra, EPE (Other); Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Sponsor-Investigator, Albino Maia, Director of Neuropsychiatry Unit, Champalimaud Foundation, Fundacao Champalimaud
Organization: Fundacao Champalimaud (Other)
Other Study IDs: BPD_DBS
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Mania; Parkinson Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation; Mania
MeSH Terms: conditions — Mania; Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DBS-induced Mania Cohort: Patients diagnosed with Parkinson's Disease (PD) who were submitted to deep brain stimulation (DBS) surgery irrespective of its target and who developed a manic episode or mixed affective state diagnosed after surgery and associated to DBS modulation, i.e., after switching on the device or changing modulation parameters.
  Interventions: Other: No Intervention / Exposure
- DBS Control Cohort: Patients diagnosed with PD who were submitted to DBS surgery irrespective of its target and who did not develop DBS-induced mania.
  Interventions: Other: No Intervention / Exposure

INTERVENTIONS:
Other: No Intervention / Exposure — No intervention / exposure since this is an observational study

SUMMARY:
Parkinson's Disease (PD) is a common and debilitating neurodegenerative disease. While medication can alleviate its symptoms, not all patients will adequately respond to medical therapy. For these cases, deep brain stimulation (DBS) has been used to improve symptoms and quality of life. Nevertheless, this approach is, in some cases, associated with incapacitating neuropsychiatric side-effects, including mood disturbances, such as DBS-induced mania. While this condition has important functional short- and long-term consequences for quality of life and prognosis, its pathophysiology is still poorly understood. In this project the investigators propose to conduct a retrospective and naturalistic study in PD patients in whom DBS stimulation resulted in mania or mixed state episode, to clarify if specific sociodemographic and clinical predictors, namely stimulation parameters and target locations, might be associated to the occurrence of this neuropsychiatric adverse event. Additionally, the investigators aim to clarify if the occurrence of DBS-induced mania results from the impact of specific stimulation parameters and/or target locations in functional connectivity networks. To explore this question, the investigators will use different neuroimaging analysis methods termed lesion topography analysis and lesion network mapping, in order to compute maps of the stimulated regions topography and the functional networks that are associated with DBS-mania, respectively. The data that will be analyzed in this project, including neuroimages, will be obtained retrospectively, by different Movement Disorders and Functional Surgery Groups in the context of Deep Brain Stimulation, and that has been collected according to their usual clinical practice.

DETAILED DESCRIPTION:
Parkinson's Disease is the second most common neurodegenerative disorder, characterized by very debilitating motor and non-motor symptoms. While medication can alleviate the impact of this disease in patient's daily life, not all patients will respond adequately to treatment, its benefits may not be long-lasting and/or incapacitating side-effects may result. For these cases, DBS has been used to improve symptoms and quality of life. Nevertheless, this approach may have clinically significant side-effects. In fact, important neuropsychiatric adverse events can occur as a result of DBS stimulation, including DBS-induced mania. This is a debilitating mood disorder, frequently associated to a decrease in DBS efficacy due to the need to change/alter stimulation parameters or switch off the device entirely with the patient losing the benefits and the improving quality of life associated with the amelioration of his motor (but also non-motor) symptoms provided by DBS-stimulation. However, reliable predictors for its occurrence are lacking and its pathophysiology is still poorly understood. In this project, the investigators aim to clarify if there are specific DBS electrode locations and/or stimulation parameters associated to development of DBS-induced Mania while additionally determining other potential sociodemographic and clinical predictors. The investigators also aim to further explore if DBS-induced mania results from the impact of specific stimulation parameters and/or target locations in functional connectivity networks.

The investigators hypothesize that specific stimulation parameters and treatment targets associated with DBS-induced mania stimulation will impact particular subcortical brain regions, alongside other clinical and sociodemographic predictors. Additionally, the investigators hypothesize that such specific pattern of stimulation will be associated to specific dysfunctional brain connectivity networks. To address these hypotheses, the investigators propose three specific aims:

1. To determine if there are specific DBS electrode location and/or stimulation parameters associated to development of DBS-induced Mania;
2. To determine if there are specific sociodemographic and/or clinical predictors for the emergence of DBS-induced Mania;
3. To explore if specific functional connectivity networks are associated to the DBS target location and/or stimulation parameters associated with Mania.

ELIGIBILITY:
DBS-induced mania cohort:

Inclusion Criteria:

* Age≥18-years-old;
* Patients diagnosed with PD who were submitted to DBS surgery irrespective of its target;
* Manic episode or mixed affective state diagnosed after surgery and associated to DBS modulation, i.e., after switching on the device or changing modulation parameters.

Exclusion Criteria:

* Patients diagnosed with bipolar disorder, or manic episode, or mixed affective state before the age of 18
* Patients diagnosed with bipolar disorder, or manic episode, or mixed affective state, before DBS surgery.

DBS Control Cohort:

A control cohort will also be collected. These patients will also meet the aforementioned inclusion and exclusion criteria with the exception of not having presented a manic episode or mixed affective state diagnosed after surgery and associated to DBS modulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be collected retrospectively from DBS surgery databases from different Movement Disorders and Functional Surgery Groups and further analyzed at the Champalimaud Neuropsychiatry Unit. Data collection will be conducted by each center independently under the approval of their respective Ethics Committees. The data that will be analyzed in this project, including neuroimages, has been collected according to the usual clinical practice of the Movement Disorders and Functional Surgery Groups.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Topographic localization of volume of tissue activation (VTA) in DBS-induced mania | From DBS parametres change until the date of first documented manic symptoms, assessed up to 24 months
  Differences in voxel-wise topographic localization of VTAs between DBS-induced mania in Parkinson's Disease (PD) and DBS PD controls. VTAs will be obtained using DBS electrodes locations and stimulation parameters.

SECONDARY OUTCOMES:
Sociodemographic and/or clinical predictors of DBS-induced mania | From DBS parametres change until the date of first documented manic symptoms, assessed up to 24 months
  Level of prediction of different models for DBS-induced mania in PD, when compared to DBS PD controls. Such models will explore different sociodemographic and/or clinical variables.
Connectivity profile of volume of tissue activation (VTA) in DBS-induced mania | From DBS parametres change until the date of first documented manic symptoms, assessed up to 24 months
  Differences in voxel-wise connectivity profile of VTAs between DBS-induced mania in PD and DBS PD controls.

CONTACTS AND LOCATIONS:
Overall Officials: Albino J. Oliveira-Maia, MD, MPH, PhD, Principal Investigator — Champalimaud Foundation
Locations (1):
- Champalimaud Foundation, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Mhyre TR, Boyd JT, Hamill RW, Maguire-Zeiss KA. Parkinson's disease. Subcell Biochem. 2012;65:389-455. doi: 10.1007/978-94-007-5416-4_16. PMID 23225012
- [Background] Nutt JG, Wooten GF. Clinical practice. Diagnosis and initial management of Parkinson's disease. N Engl J Med. 2005 Sep 8;353(10):1021-7. doi: 10.1056/NEJMcp043908. No abstract available. PMID 16148287
- [Background] Benabid AL, Pollak P, Louveau A, Henry S, de Rougemont J. Combined (thalamotomy and stimulation) stereotactic surgery of the VIM thalamic nucleus for bilateral Parkinson disease. Appl Neurophysiol. 1987;50(1-6):344-6. doi: 10.1159/000100803. PMID 3329873
- [Background] Siegfried J, Lippitz B. Bilateral chronic electrostimulation of ventroposterolateral pallidum: a new therapeutic approach for alleviating all parkinsonian symptoms. Neurosurgery. 1994 Dec;35(6):1126-9; discussion 1129-30. doi: 10.1227/00006123-199412000-00016. PMID 7885558
- [Background] Pollak P, Benabid AL, Gross C, Gao DM, Laurent A, Benazzouz A, Hoffmann D, Gentil M, Perret J. [Effects of the stimulation of the subthalamic nucleus in Parkinson disease]. Rev Neurol (Paris). 1993;149(3):175-6. French. PMID 8235208
- [Background] Deep-Brain Stimulation for Parkinson's Disease Study Group; Obeso JA, Olanow CW, Rodriguez-Oroz MC, Krack P, Kumar R, Lang AE. Deep-brain stimulation of the subthalamic nucleus or the pars interna of the globus pallidus in Parkinson's disease. N Engl J Med. 2001 Sep 27;345(13):956-63. doi: 10.1056/NEJMoa000827. PMID 11575287
- [Background] Mosley PE, Marsh R. The psychiatric and neuropsychiatric symptoms after subthalamic stimulation for Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2015 Winter;27(1):19-26. doi: 10.1176/appi.neuropsych.14040069. PMID 25716484
- [Background] Accolla EA, Pollo C. Mood Effects After Deep Brain Stimulation for Parkinson's Disease: An Update. Front Neurol. 2019 Jun 14;10:617. doi: 10.3389/fneur.2019.00617. eCollection 2019. PMID 31258509
- [Background] Mosley PE, Smith D, Coyne T, Silburn P, Breakspear M, Perry A. The site of stimulation moderates neuropsychiatric symptoms after subthalamic deep brain stimulation for Parkinson's disease. Neuroimage Clin. 2018 Mar 13;18:996-1006. doi: 10.1016/j.nicl.2018.03.009. eCollection 2018. PMID 29876284
- [Background] Boes AD, Prasad S, Liu H, Liu Q, Pascual-Leone A, Caviness VS Jr, Fox MD. Network localization of neurological symptoms from focal brain lesions. Brain. 2015 Oct;138(Pt 10):3061-75. doi: 10.1093/brain/awv228. Epub 2015 Aug 10. PMID 26264514
- [Background] Fox MD. Mapping Symptoms to Brain Networks with the Human Connectome. N Engl J Med. 2018 Dec 6;379(23):2237-2245. doi: 10.1056/NEJMra1706158. No abstract available. PMID 30575457
- [Background] Cotovio G, Talmasov D, Barahona-Correa JB, Hsu J, Senova S, Ribeiro R, Soussand L, Velosa A, Silva VCE, Rost N, Wu O, Cohen AL, Oliveira-Maia AJ, Fox MD. Mapping mania symptoms based on focal brain damage. J Clin Invest. 2020 Oct 1;130(10):5209-5222. doi: 10.1172/JCI136096. PMID 32831292
- [Background] Barahona-Correa JB, Cotovio G, Costa RM, Ribeiro R, Velosa A, Silva VCE, Sperber C, Karnath HO, Senova S, Oliveira-Maia AJ. Right-sided brain lesions predominate among patients with lesional mania: evidence from a systematic review and pooled lesion analysis. Transl Psychiatry. 2020 May 12;10(1):139. doi: 10.1038/s41398-020-0811-0. PMID 32398699
- [Background] van den Heuvel MP, Hulshoff Pol HE. Exploring the brain network: a review on resting-state fMRI functional connectivity. Eur Neuropsychopharmacol. 2010 Aug;20(8):519-34. doi: 10.1016/j.euroneuro.2010.03.008. Epub 2010 May 14. PMID 20471808
- [Background] Fox MD, Greicius M. Clinical applications of resting state functional connectivity. Front Syst Neurosci. 2010 Jun 17;4:19. doi: 10.3389/fnsys.2010.00019. eCollection 2010. PMID 20592951
- [Background] Yeo BT, Krienen FM, Sepulcre J, Sabuncu MR, Lashkari D, Hollinshead M, Roffman JL, Smoller JW, Zollei L, Polimeni JR, Fischl B, Liu H, Buckner RL. The organization of the human cerebral cortex estimated by intrinsic functional connectivity. J Neurophysiol. 2011 Sep;106(3):1125-65. doi: 10.1152/jn.00338.2011. Epub 2011 Jun 8. PMID 21653723
- [Background] Buckner R, Roffman J, Smoller J. Brain Genomics Superstruct Project (GSP). Harv Dataverse. 2014;10.
- [Background] Darby RR, Laganiere S, Pascual-Leone A, Prasad S, Fox MD. Finding the imposter: brain connectivity of lesions causing delusional misidentifications. Brain. 2017 Feb;140(2):497-507. doi: 10.1093/brain/aww288. Epub 2017 Jan 12. PMID 28082298
- [Background] Darby RR, Horn A, Cushman F, Fox MD. Lesion network localization of criminal behavior. Proc Natl Acad Sci U S A. 2018 Jan 16;115(3):601-606. doi: 10.1073/pnas.1706587115. Epub 2017 Dec 18. PMID 29255017
- [Background] Padmanabhan JL, Cooke D, Joutsa J, Siddiqi SH, Ferguson M, Darby RR, Soussand L, Horn A, Kim NY, Voss JL, Naidech AM, Brodtmann A, Egorova N, Gozzi S, Phan TG, Corbetta M, Grafman J, Fox MD. A Human Depression Circuit Derived From Focal Brain Lesions. Biol Psychiatry. 2019 Nov 15;86(10):749-758. doi: 10.1016/j.biopsych.2019.07.023. Epub 2019 Aug 2. PMID 31561861
- [Background] Eklund A, Nichols TE, Knutsson H. Cluster failure: Why fMRI inferences for spatial extent have inflated false-positive rates. Proc Natl Acad Sci U S A. 2016 Jul 12;113(28):7900-5. doi: 10.1073/pnas.1602413113. Epub 2016 Jun 28. PMID 27357684
- [Background] Poldrack RA, Baker CI, Durnez J, Gorgolewski KJ, Matthews PM, Munafo MR, Nichols TE, Poline JB, Vul E, Yarkoni T. Scanning the horizon: towards transparent and reproducible neuroimaging research. Nat Rev Neurosci. 2017 Feb;18(2):115-126. doi: 10.1038/nrn.2016.167. Epub 2017 Jan 5. PMID 28053326